CLINICAL TRIAL: NCT05260905
Title: Predictors of Affective Responses to Sprint Interval Exercise
Status: Active, not recruiting | Type: Observational
Sponsor: University of Stirling (Other)
Collaborators: Swansea University (Other); University of Worcester (Other); University of Edinburgh (Other); California State University, San Marcos (Other)
Responsible Party: Principal Investigator, Niels Vollaard, Principal investigator, University of Stirling
Other Study IDs: NICR4297
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: General Health
Keywords: Affective valence; Affect; REHIT; Reduced-exertion high-intensity interval training

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: All participants will perform 2 experimental sessions, each involving a REHIT exercise session.
  Interventions: Behavioral: REHIT

INTERVENTIONS:
Behavioral: REHIT — REHIt involves 10 minutes of unloaded cycling on a stationary bike, interspersed with two 20-s 'all-out' cycle sprints against a resistance equivalent to 7.5% of body mass.
  Other Names: Reduced-exertion high-intensity interval training

SUMMARY:
Regular exercise is needed to ensure good general health and wellbeing. How exercise makes you feel (pleasant / unpleasant) is thought to be important for whether people will stick with a given exercise routine. Sprint interval training (SIT) has been shown be a time-efficient exercise strategy for improving health, but some researchers suggest that SIT may be experienced as unpleasant and therefore unsuitable as an exercise routine for improving general health and wellbeing. However, SIT protocols are diverse, and it has previously been shown that very short SIT protocols such as 'reduced-exertion high-intensity interval training' (REHIT) are not perceived as unpleasant, at least on average. Interestingly, how REHIT is perceived appears to be highly variable between individuals. This individual variability may have important implications for whether people stick with REHIT and/or SIT in real-world settings, and therefore it is important to characterise it and better understand why some people find this exercise unpleasant while others do not. This study aims to characterise the within-participant and between-participant variability in how people perceive REHIT. Furthermore, potential relationships between psychological characteristics and how people perceive REHIT will be explored.

DETAILED DESCRIPTION:
The study will recruit between 100-150 apparently healthy participants from multiple sites. Participants will be asked to complete the following questionnaires: Anxiety Sensitivity Index 3 (ASI-3), Body Perception Questionnaire (BPQ), Sense of Agency Scale (SoAS), and Preferences and Tolerances for High Intensity Exercise (PRETIE-Q). This data will be used to determine if changes in affective valence during REHIT are associated with the responses to these questionnaires.

Participants' maximal aerobic capacity (VO2max) will be determined using an incremental cycling test to exhaustion. Participants will start cycling on a stationary bike at a low intensity (30 W). The intensity will increase by 1 W every 3 seconds until volitional exhaustion or an inability to maintain a pedalling frequency of >60 rpm. Expired O2 and CO2 will be continuously measured breath-by-breath using an online gas analyser. VO2max will be determined as the highest value for a 15-breath rolling average of VO2. VO2max will be accepted if at least 2 of the following criteria are met: volitional exhaustion, inability to maintain a pedal frequency of 60 rpm, RER>1.10, a plateau in VO2, and/or heart rate within 10 bpm of the age predicted maximum (220-age).

Participants will practice REHIT exercise on 2 occasions. Each session will be performed on a mechanically-braked cycle ergometer. REHIT consists of 10 minutes of unloaded cycling interjected with 2 maximal sprints against a resistance equivalent to 7.5% baseline body mass. In the first practice session the sprints will be 10 seconds long; in the second practice session they will be 15 seconds long. Sprints will finish at 2 minutes and 6 minutes into the session. The scales for rating of perceived exertion (RPE, Borg scale), affect (Feeling scale), and arousal (Felt Arousal) will be explained to the participants during the familiarisation sessions.

The final 2 sessions are the experimental sessions and will involve REHIT sessions with 20-second sprints. The Demand and Resource Questionnaire will be administered pre-exercise. Affect (Feeling scale) and arousal (Felt Arousal) will be measured at rest before exercise and at the end of every minute during exercise. Rating of perceived exertion (RPE, Borg scale) will be measured at the same time-points but during exercise only. Heart rate and power output will be measured throughout the 10-minute exercise session. The Physical Activity Enjoyment Scale (PACES) will be administered 10 minutes after exercise.

Within- and between-participant variability in the change in affect with exercise will be determined. Potential associations between psychology questionnaire scores and the change in affect with exercise will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy
* Sedentary or recreationally active

Exclusion Criteria:

* Classified as highly physically active on the International Physical Activity Questionnaire (IPAQ)
* Answering 'Yes' to any of the questions of a standard Physical Activity Readiness Questionnaire (PAR-Q)
* Resting heart rate >100 bpm
* Resting blood pressure > 140/90 mm Hg
* BMI > 35 kg/m2
* Testing positive for Covid-19
* Pregnant women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of any apparently healthy individuals who are not highly physically active and who have no contra-indications to performing exercise.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Exercise-induced change in affective valence | Affective valence will be measured before exercise and at the end of every minute during the 10-minute exercise trials. The outcome measure will be determined as the differences between the pre-exercise measurement and the lowest value during exercise.
  Affective valence is a measure of how pleasant / unpleasant the exercise is and will be measured using the 11-point Feeling Scale pre-exercise (ranging from 5 (very bad) to 5 (very good)), and at the end of every minute during exercise. The change in affect will be calculated as the difference between the pre-exercise value and the lowest value during exercise. This will be measured during both experimental sessions.

SECONDARY OUTCOMES:
Rating of perceived exertion (RPE) | RPE will be measured at the end of every minute during the 10-minute exercise trials.
  RPE is a measure of how hard an exercise session is perceived to be and will be measured using the 15-point Borg scale (ranging from 6 (very very light) to 20 (very very hard) at the end of every minute during exercise. RPE will be measured during both experimental sessions.
Felt arousal | Felt arousal will be measured at the end of every minute during the 10-minute exercise trials.
  Felt arousal is a measure of perceived activation and will be measured using the Felt Arousal Scale (FAS) along a 6-point scale (ranging from low arousal (1) to high arousal (6)), at the end of every minute during exercise. Felt arousal will be measured during both experimental sessions.

OTHER OUTCOMES:
Body awareness and autonomic reactivity | Body awareness and autonomic reactivity will be measured at the start of the study before any exercise sessions are performed.
  Body awareness and autonomic reactivity will be measured using the Body Perception Questionnaire (BPQ), with scores ranging from 26 (poor body awareness and autonomic reactivity) to 118 (excellent body awareness and autonomic reactivity).
Anxiety sensitivity | Anxiety sensitivity will be measured at the start of the study before any exercise sessions are performed.
  Anxiety sensitivity measures concern associated with possible negative consequences of anxiety-related symptoms and is assessed using the Anxiety Sensitivity Index-3 (ASI-3) on a scale from 0 (almost no anxiety sensitivity) to 72 (high anxiety sensitivity).
Preference for and tolerance of the intensity of exercise | Preference for and tolerance of the intensity of exercise will be measured at the start of the study before any exercise sessions are performed.
  Preference for and tolerance of the intensity of exercise will be assessed using the PRETIE-Q questionnaire. Preference for the intensity of exercise is measured on a scale from 8 (low) to 40 (high) and tolerance of the intensity of exercise is measured on a scale from 8 (low) to 40 (high).
Sense of agency | Sense of agency will be measured at the start of the study before any exercise sessions are performed.
  Sense of agency is a measure of to what extent someone feels they are the initiator of their own actions, and will will be assessed using the Sense of Agency Scale (SoAS) on a scale of 13 (low sense of agency) to 91 (high sense of agency).
Exercise enjoyment | Exercise enjoyment will be measured 10 minutes after the final experimental exercise session.
  Exercise enjoyment will be measured using the Physical Activity Enjoyment Scale (PACES), on a scale from 0 (no enjoyment) to 48 (very high enjoyment).
Exercise power output | Power output will be measured continuously during each of the 2 20-second cycle sprints in the exercise trials.
  Power output during the 'all-out' cycle sprints will be measured, and quantified as the peak power output (in Watts), mean power output (in Watts), and fatigue index (drop in power from highest to lowest, expressed as a percentage of peak power output).
Self efficacy to do exercise | Self efficacy will be measured directly before each of the two experimental trials.
  Self efficacy will be assessed using the Demand and Resource Questionnaire, which assesses how demanding the participants consider the upcoming exercise to be (on a scale from 1 (not at all) to 6 (extremely)), and how well they think they will cope with these demands (on a scale from 1 (not at all) to 6 (extremely)).

CONTACTS AND LOCATIONS:
Overall Officials: Niels Vollaard, PhD, Principal Investigator — University of Stirling
Locations (1):
- University of Stirling, Stirling, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised IPD can be provided to other researchers on request, if the data are of use to answer a valid research question.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of data collection.
Access Criteria: Academic researchers aiming to answer a valid research question.